CLINICAL TRIAL: NCT07396610
Title: Comparative Evaluation of a Bioactive Glass Dentifrice and 810 nm Diode Laser for Dentinal Hypersensitivity: A Randomized Placebo-Controlled Clinical Study
Brief Title: Effect of Diode Laser and Bioactive Glass on Dentinal Hypersensitivity
Acronym: Laser & Bioact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Professor, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRGCDS/2024/044; RGP1/3/46 (Other Grant/Funding Number: The Deanship of Scientific Research at King Khalid University)
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dentinal Hypersensitivity
Keywords: Dentinal Hypersensitivity; Diode Laser; 810-nm Diode Laser; Bioactive Glass; Desensitizing Agents
MeSH Terms: interventions — Lasers, Semiconductor; NovaMin

STUDY DESIGN:
Intervention Model Description: Participants with dentinal hypersensitivity are randomly assigned to one of three parallel groups to receive either 810-nm diode laser therapy, a bioactive glass-based desensitizing agent, or a placebo intervention. Each participant receives only the assigned intervention and is followed longitudinally for outcome assessment.
Who Masked: Participant
Masking Description: Participants are blinded to the assigned intervention. The diode laser, bioactive glass application, and placebo procedures are designed to appear similar to participants to minimize expectation bias. Outcome assessments are conducted using standardized protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diode Laser Group (Experimental): Participants receive 810-nm diode laser therapy applied to hypersensitive dentin.
  Interventions: Device: 810-nm Diode Laser
- Bioactive Glass Group (Experimental): Participants receive a bioactive glass-based desensitizing agent applied to hypersensitive dentin
  Interventions: Drug: Bioactive Glass (NovaMin)
- Placebo Group (Placebo Comparator): Participants receive a placebo intervention without active desensitizing properties.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: 810-nm Diode Laser — Non-contact diode laser irradiation applied to exposed dentin
  Arms: Diode Laser Group
Drug: Bioactive Glass (NovaMin) — Topical application of bioactive glass-containing desensitizing agent
  Arms: Bioactive Glass Group
Other: Placebo — Inactive material resembling test interventions.
  Arms: Placebo Group

SUMMARY:
Dentinal hypersensitivity is a common clinical condition characterized by short, sharp pain arising from exposed dentin in response to thermal, tactile, or evaporative stimuli. It can significantly affect oral health-related quality of life and routine dental care. Various treatment approaches have been proposed, including laser therapy and bioactive materials, with differing mechanisms of action and clinical outcomes.

This randomized controlled clinical trial aims to compare the effectiveness of an 810-nm diode laser, a bioactive glass-based desensitizing agent, and a placebo in reducing dentinal hypersensitivity. Eligible participants with clinically diagnosed dentinal hypersensitivity will be randomly assigned to one of three parallel treatment groups. Pain intensity will be assessed using a visual analog scale following standardized air stimulus testing at baseline and at predefined follow-up intervals.

The study will evaluate both immediate and long-term changes in hypersensitivity over a 12-month follow-up period. The findings are intended to provide clinical evidence on the comparative performance of diode laser therapy and bioactive glass in the management of dentinal hypersensitivity.

DETAILED DESCRIPTION:
Dentinal hypersensitivity is a frequently encountered clinical condition characterized by a short, sharp pain arising from exposed dentin in response to thermal, tactile, osmotic, or evaporative stimuli. The condition is commonly associated with gingival recession, enamel loss, or dentin exposure due to abrasion, erosion, or periodontal therapy. Despite its high prevalence, the management of dentinal hypersensitivity remains challenging, and no single treatment approach has been universally accepted as the gold standard.

Conventional management strategies are primarily based on either neural desensitization or occlusion of dentinal tubules. Bioactive glass-based desensitizing agents, such as those containing calcium sodium phosphosilicate, act by releasing calcium and phosphate ions that form a hydroxycarbonate apatite-like layer, leading to physical occlusion of dentinal tubules. In contrast, diode laser therapy has been proposed to reduce dentinal hypersensitivity through mechanisms that may include alteration of nerve conduction, coagulation of dentinal proteins, and partial sealing of dentinal tubules. However, the comparative clinical effectiveness and durability of these treatment modalities remain unclear, particularly over long-term follow-up periods.

This randomized controlled clinical trial is designed to compare the effects of an 810-nm diode laser, a bioactive glass-based desensitizing agent, and a placebo intervention in the management of dentinal hypersensitivity. Eligible participants diagnosed with dentinal hypersensitivity based on clinical examination and positive response to standardized air stimulus testing will be randomly allocated into three parallel treatment groups. Randomization will be performed using an appropriate allocation method to ensure balanced group distribution.

Participants in the diode laser group will receive non-contact laser irradiation applied to exposed dentin surfaces using an 810-nm diode laser at a standardized power setting and exposure duration. Participants in the bioactive glass group will receive topical application of a bioactive glass-containing desensitizing agent according to manufacturer-recommended instructions. The placebo group will receive an inactive intervention designed to mimic the appearance and application procedure of the active treatments without containing therapeutic components.

Pain intensity will be assessed using a visual analog scale following standardized air stimulus testing. Outcome assessments will be conducted at baseline, immediately after treatment, and during follow-up visits at 1 month, 6 months, and 12 months. The primary outcome measure will be the change in dentinal hypersensitivity pain scores from baseline. Secondary outcomes will include the sustainability of pain reduction and participant-reported comfort over time.

All clinical procedures and assessments will be performed by trained personnel following standardized protocols to minimize variability. Ethical approval will be obtained from the appropriate institutional review board or ethics committee prior to study initiation, and written informed consent will be obtained from all participants. The results of this study are intended to provide clinically relevant evidence regarding the comparative performance of diode laser therapy and bioactive glass-based desensitizing agents for the management of dentinal hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years
* Presence of clinically diagnosed dentinal hypersensitivity in at least one tooth
* Positive response to standardized air stimulus test
* Good general and oral health

Exclusion Criteria:

* Presence of dental caries, defective restorations, or cracked teeth in the study tooth
* Evidence of pulpal pathology or periapical disease
* Periodontal disease requiring active treatment
* Use of desensitizing agents or sensitivity treatments within the previous 4 weeks
* History of allergy or hypersensitivity to any study materials
* Systemic conditions or medications that may affect pain perception
* Pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Dentinal Hypersensitivity Pain Score | Baseline, immediately after treatment, 1 month, 6 months, and 12 months
  Change in pain intensity associated with dentinal hypersensitivity measured using a visual analog scale (VAS) following standardized air stimulus testing on the affected tooth.

SECONDARY OUTCOMES:
Sustained Reduction in Dentinal Hypersensitivity | 6 months and 12 months
  Assessment of long-term changes in dentinal hypersensitivity pain scores measured using a visual analog scale (VAS) following standardized air stimulus testing.
Participant-Reported Comfort Level | 1 month and 6 months
  Participant-reported perception of comfort and sensitivity related to the treated tooth, recorded using a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sri Rajiv Gandhi College of Dental Sciences & Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. The dataset contains sensitive clinical and personal information, and participant consent does not include provisions for public data sharing. De-identified aggregate data will be reported through publications and trial registry results in accordance with ethical approvals and institutional policies.